CLINICAL TRIAL: NCT01158781
Title: Restoration of Life Role Participation Through Integrated Cognitive and Motor Training for Individuals With TBI
Brief Title: Restoration of Life Role Participation Through Cognitive and Motor Training for TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malcom Randall VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janis Daly, Director, Brain Rehabilitation Research Center, North Florida/South Georgia Veterans Health System
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PT074749
Record Dates: First submitted 2009-10-13; First posted 2010-07-08 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; motor learning; robotics; Functional electrical stimulation
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gait, balance, arm function, cognition (Experimental): 12 weeks of training for balance, gait, upper limb function, and cognition
  Interventions: Behavioral: Experimental: gait, balance, arm function, cognition

INTERVENTIONS:
Behavioral: Experimental: gait, balance, arm function, cognition — 12 weeks of training for balance, gait, upper limb function, and cognition, including functional electrical stimulation with surface electrodes, robotics, and motor learning

SUMMARY:
The purpose of this study is to restore life role participation for those with TBI by customizing, applying, and testing integrated cognitive and motor training protocols that were successful in populations with impairments similar to TBI. The treatment protocols are based on principles of brain plasticity and re-learning, required to restore cognitive and motor function. The intervention targets an array of impairments that are obstacles to life role participation. These include cognitive attention and executive control; motor control for upper limb function; balance and gait; and cognitive executive control of simultaneous cognitive and motor tasks required by everyday tasks. The intervention utilizes training specificity, framing the intervention within functional task and life role activity component practice.

DETAILED DESCRIPTION:
The investigators will use an assessment and treatment decision schema that has been successful in restoration of life role participation for stroke survivors and a comparable schema used for cognitive training for TBI patients. The subject assessment and decision schema will be used to identify for each subject, the optimal array of impairment interventions. The proposed treatment will optimize outcome by customizing the intervention and use of technologies, while ensuring the application of the array of impairment interventions required to produce restoration of function and life role participation. The investigators will target an array of impairments preventing participation in life role activities, which will include dyscoordination and weakness of upper limb, impaired balance, gait deficits, and impaired attention and executive function. In treatment, the investigators will use a dual-task paradigm combining motor and cognitive training, with treatment extending to the every day environment. Treatment will be up to 5 times/wk, 5hrs/day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Medically Stable
* Age > 18 years
* Ability to walk at least with the minimum assistance of one person or an assistive device
* At least 6 months post injury
* Ability to follow 2 stage commands

Exclusion Criteria:

* pacemaker
* Acute medical conditions
* potential subjects will undergo a screening evaluation to determine eligibility for study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-05; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Berg Balance | week 12
  Balance function

CONTACTS AND LOCATIONS:
Overall Officials: Janis Daly, Ph.D., M.S., Principal Investigator — US Department of Veterans Affairs
Locations (1):
- Gainesville VA Medical Center, Gainesville, Florida, United States